CLINICAL TRIAL: NCT06253026
Title: Physiological, Psychological and Cognitive Impact of Air Search and Rescue Missions
Brief Title: Fatigue in Air Search and Rescue Missions
Status: Recruiting | Type: Observational
Sponsor: Faculdade de Motricidade Humana (Other)
Collaborators: CIDEFES - Universidade Lusofona (Unknown); Força Aerea Portuguesa (Unknown)
Responsible Party: Sponsor
Other Study IDs: LabFisiolBioqFAP
Record Dates: First submitted 2023-12-21; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Fatigue Syndrome, Chronic
Keywords: Fatigue; Strength; Sleep pattern; Cognition
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum for biochemical analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Air mission personnel: Military crew that goes to air search and rescue missions in groups of five
  Interventions: Other: Search and rescue mission
- Control: Ground military personnel

INTERVENTIONS:
Other: Search and rescue mission — Air search and rescue missions lasting 15 consecutive days
  Groups: Air mission personnel

SUMMARY:
The purpose of this observational study is to understand and evaluate the physiological, psychological, and cognitive impact of 15 consecutive days of air search and rescue mission deployments on Portuguese Air Force crews. The main goals are: 1) Characterize and compare the body composition, cardiorespiratory fitness, and strength levels of air force search and rescue mission crew members with different tasks; 2) Characterize the physiological, psychological and cognitive impacts induced by a single deployment; 3) Identify possible cumulative effects of successive deployments on the variables of interest; 3) Characterize the changes in lifestyle, quality of sleep and nutrition induced by the deployments. The participants will be evaluated after a period of hollidays, before missions, during missions, upon arrival, for a period of twelve months, and at the end of twelve months.

DETAILED DESCRIPTION:
Fatigue, especially in its mental and physical forms, impacts aviation performance and can result from sleep deprivation, prolonged wakefulness, changes in the circadian cycle and eating patterns, or excessive workload. The Air Force's multidisciplinary teams deployed to complex missions, where physical and mental demands are known to be different between each operational element, face the need for diligence and efficiency to avoid errors that could result in fatal consequences. Physical and mental recovery becomes crucial for optimal performance in missions that require precision, physical robustness and mental acuity. Furthermore, fatigue can have long-term health effects, associated with reduced work capacity and possibly depression and anxiety. Understanding the physiological and psychological impact of each mission highlights the need for corrective and preventative measures to increase success and safety. The objective of the present study is to understand and evaluate the physiological, psychological and cognitive impacts after deployment missions on Portuguese Air Force personnel. Both ground personnel and air search and rescue mission crews will be evaluated after a period of holidays (baseline). During twelve months, when participants are recruited for missions, assessments will occur at three points: pre-mission, during the mission and post-mission. Twelve months after the first assessment (final), all personnel will be evaluated again. Pre-mission assessments will take place during the week prior to departure for the mission. Baseline, final and pre-mission assessments will include anthropometric measurements, assessment of body composition and water compartments, cardiorespiratory, balance and strength tests, cognitive performance, well-being, sleep quality, food intake, psychological tests, and blood biochemical analyses. During the mission, food intake and sleep quality will be monitored. The post-mission assessment that will be carried out upon arrival will only include water compartment assessment, strength tests, cognitive performance, well-being, psychological tests, and blood biochemical analysis. Statistical analysis will be performed using IBM SPSS Statistics software (version 28.0, NY, IBM). Descriptive analyzes will be carried out to characterize the sample. Normality for each variable of interest will be tested with the Kolmogorov-Smirnov test. Either the paired t test or the Wilcoxon test will be used to assess the effect of each 15-day mission (pre vs post). ANOVA for repeated measures (2x2) will be used to assess the cumulative effect of the missions (baseline vs final and ground personnel vs air personnel). A statistical significance of α = p<0.05 will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Air Force Military

For intervention group

* Approved for search and rescue missions by the clinical staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Military crews composed by pilot, co-pilot, nurse, host-operator, rescue diver. Land military personal involved in desk tasks.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change of Well-being Index | Every 15 days search and rescue mission, up to 1 year
  Numeric scale (0-28). A lower score is associated with a better result
Changes in response inhibition (go/no go test) | Every 15 days search and rescue mission, up to 1 year
  Number of errors, reaction time (ms)
Change in response inhibition (Stroop test) | Every 15 days search and rescue mission, up to 1 year
  Number of errors, reaction time (ms)
Change of heart rate variability | Every 15 days search and rescue mission, up to 1 year
  bpm, rr interval
Change of double task ability | Every 15 days search and rescue mission, up to 1 year
  walking and calculating
Change of maximal voluntary strength | Every 15 days search and rescue mission, up to 1 year
  N
Change of maximal Hand Grip strength | Every 15 days search and rescue mission, up to 1 year
  N
Peak tork of extensors and flexors of the tight | Every 15 days search and rescue mission, up to 1 year
  Peak tork
Isometric mid-tight pull | Every 15 days search and rescue mission, up to 1 year
  maximal tork
VO2max | 1 year
  Indirect calorimetry (mL/kg/min)
Hematological indicators (hematocrit) | Every 15 days search and rescue mission, up to 1 year
  Percentage (volume/volume) of red blood cell in total blood
Hematological indicators (hemoglobin) | Every 15 days search and rescue mission, up to 1 year
  grams/mL blood
Hematological indicators (cell counts) | Every 15 days search and rescue mission, up to 1 year
  Number of red and white cells per mL of total blood
Possible perturbations diagnosis | 1 year
  Psychology clinical interview

SECONDARY OUTCOMES:
Change in body mass BIA | Every 15 days search and rescue mission, up to 1 year
  body mass (kg)
Change in fat-free mass BIA | Every 15 days search and rescue mission, up to 1 year
  Fat-free mass (kg)
Change in fat mass BIA | Every 15 days search and rescue mission, up to 1 year
  Fat mass (kg)
Change in total water BIA | Every 15 days search and rescue mission, up to 1 year
  Total water (kg)
Change in intracellular water BIA | Every 15 days search and rescue mission, up to 1 year
  Intracellular water (kg), extracellular water (kg)
Change in extracellular water BIA | Every 15 days search and rescue mission, up to 1 year
  Extracellular water (kg)
Change in center of pressure | Every 15 days search and rescue mission, up to 1 year
  cm
Change in sleep pattern, and sleep efficiency and quality of sleep | Every 15 days search and rescue mission, up to 1 year
  Sleep minutes and minutes to fall asleep
Bone mineral content dxa | 1 year
  kg
Change in eating pattern (record) calories and macros | Every 15 days search and rescue mission, up to 1 year
  kcal/d

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Human Kinetics, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No